CLINICAL TRIAL: NCT05943184
Title: Clinical Value of Cognitive Behavioral Nursing Model to Patients With Congenital Glaucoma
Brief Title: Cognitive Behavioral Nursing Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taiyuan Central Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Yanfang Ma, Principal investigator, Taiyuan Central Hospital of Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TaiyuanCH 001
Record Dates: First submitted 2023-06-14; First posted 2023-07-13 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Behavioral Nursing; Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- Observation group (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Nursing Model

INTERVENTIONS:
Behavioral: Cognitive Behavioral Nursing Model — (1)Psychological intervention was accessible to those who felt resistant to their treatment plans or developed inferior feelings due to visual impairment to establish a good relationship with patients and help them better cope with unhealthy emotions. (2) Health education was provided through self-developed booklets and question-and-answer sessions to publicize the fundamental knowledge and make sure all patients have a full understanding of the disease and related treatments. (3) Dietary guidelines were set out to encourage a light, healthy diet with fruits and vegetables, free of irritating food, and containing a limited amount of oily food. (4) Behavioral guidelines were developed to address the importance of quitting tobacco use and prevent eye strain due to excessive eye use with tailored eye care plans.
  Arms: Observation group

SUMMARY:
Materials and Methods

1. General information This study enrolled 153 patients with congenital glaucoma who were treated at our hospital from January 2021 to December 2022. These patients were divided into an observation group (n = 76) and a control group (n = 77) using a random number table. The inclusion criteria were as follows: (1) meeting the diagnostic criteria for glaucoma, (2) following the attending doctor's recommendations to receive surgical treatment, and (3) volunteering to participate in the study. The exclusion criteria were as follows: (1) severe organic dysfunction, (2) cardiovascular and/or cerebrovascular diseases, (3) hypertension, (4) contraindications for surgery, (5) other eye diseases, (6) communication disorders, and (7) mental illnesses. Informed consent with signature was obtained from every participant, and the study has been approved by the hospital's ethics committee.
2. Research methods The control group was provided with routine care, including warm reception and provision of a quiet, clean, and well-ventilated ward environment for good rest. Patients were educated to broaden their knowledge of the disease and related surgical treatment, particularly the importance and outcomes of surgical treatment, thereby allaying their feeling of fear and boosting their confidence in recovery. Meanwhile, patients were encouraged to break their unhealthy habits, avoid bad diet choices, and take medications on time.

   The observation group received CBNI described as follows: (1) A cognitive-behavioral intervention group was set up by several nurses who had a background of systematic cognitive intervention training, were able to independently develop comprehensive behavioral intervention plans and assess a patient's cognitive level, and had an adequate understanding of the fundamentals of cognitive behavioral intervention. Through thorough communication with patients, these nurses were supposed to identify their major concerns and assess their cognitive behavior. Based on the assessment results, psychological counseling was provided for every patient, with each session lasting at least 50 minutes. In addition, the nurses were required to reassure all patients by proactively introducing the precautions of surgery and nursing care. (2) Psychological intervention was accessible to those who felt resistant to their treatment plans or developed inferior feelings due to visual impairment to establish a good relationship with patients and help them better cope with unhealthy emotions. Professional education was provided through communication with patients so that they could gain detailed knowledge of the disease. Chatting and music were useful to relieve tension and psychological stress. Regular patient support groups were organized to help patients develop confidence and a positive attitude toward the disease. (3) Health education was provided through self-developed booklets and question-and-answer sessions to publicize the fundamental knowledge and make sure all patients have a full understanding of the disease and related treatments. The nurses were also required to closely monitor patient compliance from the perspectives of diet, lifestyle, psychology, and treatment. (4) Dietary guidelines were set out to encourage a light, healthy diet with fruits and vegetables, free of irritating food, and containing a limited amount of oily food. It should be noted that smooth bowel movements are essential to prevent increased IOP induced by constipation. Therefore, the recommended diet is high in dietary fiber and fruits. (5) Behavioral guidelines were developed to address the importance of quitting tobacco use and prevent eye strain due to excessive eye use with tailored eye care plans. The nurses were responsible for guiding the proper use of eye drops by patients, reminding all patients to seek medical attention immediately if they experienced any eye discomfort, and stressing the risk of increasing IOP due to prolonged periods of looking down and other unhealthy habits.
3. Statistical analysis The software SPSS22.0 was used for data analysis. Measurement data were expressed as "mean ± standard deviation (x±s)", and comparisons between the two groups were examined by the t-test. Enumeration data were represented as percentages (%) and inter-group comparisons were examined using the χ2 test. Significance was set at the level of P <0.05.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnostic criteria for glaucoma;
* following the attending doctor's recommendations to receive surgical treatment, and;
* volunteering to participate in the study

Exclusion Criteria:

* severe organic dysfunction;
* cardiovascular and/or cerebrovascular diseases;
* hypertension;
* contraindications for surgery;
* other eye diseases;
* communication disorders;
* mental illnesses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
SDS scores | before and at one month of nursing intervention
  The cutoff score for SAS is 50, with scores of 50-59 indicative of mild anxiety, 60-69 of moderate anxiety, and scores above 70 of severe anxiety.
SAS scores | before and at one month of nursing intervention
  The cutoff score for SDS is 53, with scores of 53-62 standing for mild depression, 63-72 for moderate depression, and scores above 72 for severe depression.
Psychological resilience | Baseline (Before the intervention)
  The level of psychological resilience was evaluated using the Connor-Davidson Resilience Scale, which covers three dimensions: optimism, self-efficacy, and resilience, with the total score ranging from 0 to 100, and higher scores reflecting greater resilience.
Patient compliance | Immediately after nursing
  The level of patient compliance during the perioperative period was assessed using an evaluation form that describes the level of compliance as complete compliance (compliance with all medical orders, surgical procedures, dietary guidelines, and schedule), partial compliance (occasional compliance with all medical orders, surgical procedures, dietary guidelines, and schedule), or noncompliance (failure to meet any of the above-mentioned criteria). The compliance rate (%) was calculated as (complete compliance + partial compliance) / total cases × 100%.
Visual acuity (VA) | At 2 weeks of nursing intervention
  a higher VA value indicates better treatment outcomes
IOP | At 2 weeks of nursing intervention
  a lower IOP values indicates better treatment outcomes
mean deviation (MD) | At 2 weeks of nursing intervention
  a lower MD values indicates better treatment outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Taiyuan Central hospital of Shanxi Medical University, Taiyuan, Shanxi, China